CLINICAL TRIAL: NCT04709328
Title: An Adaptive, Randomized, Double-blinded, Placebo-controlled Phase II/III Trial of Monoclonal Antibody SCTA01 Against SARS-CoV-2 in High-Risk Outpatients With COVID-19 (MAOP3 Trial)
Brief Title: To Evaluate SCTA01 Treatment of High-risk Outpatients With COVID-19
Acronym: MAOP3
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCTA01-A301
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — upanovimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SCTA01 low dose +SOC (Experimental): SCTA01, a recombinant anti-SARS-CoV-2 spike protein monoclonal antibody
  Interventions: Drug: SCTA01
- SCTA01 middle dose+SOC (Experimental): SCTA01, a recombinant anti-SARS-CoV-2 spike protein monoclonal antibody
  Interventions: Drug: SCTA01
- SCTA01 High dose +SOC (Experimental): SCTA01, a recombinant anti-SARS-CoV-2 spike protein monoclonal antibody
  Interventions: Drug: SCTA01
- Placebo+SOC (Placebo Comparator): SCTA01, a recombinant anti-SARS-CoV-2 spike protein monoclonal antibody
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SCTA01 — Diluted by 0.9% normal saline，IV
  Arms: SCTA01 High dose +SOC; SCTA01 low dose +SOC; SCTA01 middle dose+SOC
Other: Placebo — IV
  Arms: Placebo+SOC

SUMMARY:
The study is a multicenter, adaptive, randomized, double-blinded and placebo-controlled Phase II/III clinical trial. It will be conducted at selected investigational sites globally. The study is comprised of 2 parts.

DETAILED DESCRIPTION:
The study is a multicenter, adaptive, randomized, double-blinded, and placebocontrolled Phase II/III trial. It will be conducted globally. The study will evaluate the efficacy and safety of SCTA01 in high-risk outpatients with COVID-19.The primary objective of the study is to evaluate the clinical efficacy rate among study group [SCTA01+ standard of care (SOC)] and control group (placebo + SOC) up to Day 29.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female adults, ≥18 years old of age at the time of randomization;
* Participants should have at least one of COVID-19 risk factor;
* Participants should have at least 2 COVID-19 related symptoms;
* Has symptoms consistent with COVID-19 as determined by the investigator with onset ≤7 days before randomization;
* First positive SARS-CoV-2 viral infection tested (PCR or antigen-based diagnostic tests) in samples collected ≤3 days prior to start of the infusion;
* Participants are currently not hospitalized;
* Participant (or legal authorized representative) has signed the ICF before any clinical activity related to SCTA01 trial;
* Women with childbearing potential must agree to use effective contraceptive methods during the study period;
* Patient should not participate in other clinical studies related to COVID-19 or SARS-CoV-2 infection.

Exclusion Criteria:

* Have known allergies to any of the components used in the formulation of the SCTA01/placebo;
* Participants with a history of severe anaphylaxis, such as severe anaphylactic reaction, urticaria, and angioedema;
* Have SpO2 ≤ 93% on room air at sea level or PaO2/FiO2 < 300, respiratory rate ≥30 per minute, heart rate ≥125 per minute (FDA);
* Require mechanical ventilation or anticipated impending need for mechanical ventilation;
* Suspected or proven serious bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking part in this study;
* Have any serious concomitant systemic disease, condition or disorder that, in the opinion of the investigator, should preclude participation in this study;
* Have any co-morbidity requiring surgery within <29 days, or that is considered life threatening within 29 days;
* Have a history of previous SARS-CoV-2 infection;
* Received convalescent plasma, COVID-19 vaccine, or anti-SARS-CoV-2 spike(S) protein targeted therapy;
* Have participated in a clinical study involving an investigational intervention within past 30 days or 5-half lives of investigational product, whichever is longer;
* Have received an investigational intervention for SARS-CoV-2 prophylaxis within 30 days before dosing;
* Pregnant or lactating women;
* Anticipated hospitalization or transfer to another medical site which is not a study site within 72 hours;
* Participants unable to follow the protocol during the study;
* Participants deemed inappropriate for enrollment by the investigator due to other factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2021-03-28 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who experience COVID-19 related hospitalization (defined as at least 24 hours of acute care) or death (all cause) up to Day 29. | Day 29

SECONDARY OUTCOMES:
Time to sustained resolution of all COVID-19-related symptoms | Day 29
- Change in symptom score (total of ratings) | Day 3, 5, 7, 11, 15, 22, and 29
Time to symptom improvement; | Day 29
Proportion of participants admitted to hospital due to COVID-19 | Day 29
Proportion of participants with ≥1 COVID-19 related hospitalization | Day 29
Proportion of participants with ≥2 COVID-19 related hospitalizations | Day 29
Total number of COVID-19 related hospitalization | Day 29
Proportion of participants who experience COVID-19 related emergency room (ER) visit | Day 29
Proportion of participants with ≥1 ER visit due to COVID-19 | Day 29
Proportion of participants with ≥2 ER visits due to COVID-19 through Day 29 | Day 29
Proportion of participants admitted to an intensive care unit (ICU) due to COVID-19 | Day 29
Proportion of patients with all-cause mortality | Day 29
Proportion of participants with O2 requirement | Day 29
Proportion of participants with ventilation requirements | Day 29
Proportion of participants that achieve SARS-CoV-2 clearance in nasopharyngeal (NP) or oropharyngeal (OP) samples | Day 8, Day 15
Change from baseline (Day 1) to Day 8 or Day 15 in SARS-CoV-2 viral shedding as measured by quantitative reverse transcription polymerase chain reaction (RT-qPCR) in NP or OP samples for SARS-CoV-2 test. | Day 8, Day 15
Cumulative incidence of serious adverse events (SAEs) | Day 120
Cumulative incidence of Grade 1, 2, 3 and 4 adverse events (AEs) | Day 120
Discontinuation or temporary suspension of infusions (for any reason) | Day 120
Number and proportion of patients with ADE | Day 120
Mean concentration-time profiles of SCTA01 | Day 29
Incidence and titers (if applicable) of anti-drug antibodies (ADA) to SCTA01 | Day 1, Day 8, Day 29, and Day 120)

REFERENCES:
- [Derived] Diaz J, Fonseca A, Yan L, Liu D, Xie L. Efficacy and safety of SARS-CoV-2 neutralizing antibody, SCTA01, in high-risk outpatients diagnosed with COVID-19: A Phase II clinical trial. Contemp Clin Trials Commun. 2025 May 17;45:101496. doi: 10.1016/j.conctc.2025.101496. eCollection 2025 Jun. PMID 40520909
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343